CLINICAL TRIAL: NCT00468182
Title: Modulation of Plasmacytoid Dendritic Cell Function in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Konstantin Balashov, Associate Professor, Rutgers, The State University of New Jersey
Other Study IDs: 0220060228
Record Dates: First submitted 2007-04-30; First posted 2007-05-02 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Interferon beta; plasmacytoid dendritic cells
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1b

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: MS patients or patients with CIS (Clinically isolated syndrome) who decided to be treated with IFN-beta for 3 months (with the option to continue Rx)
  Interventions: Drug: Interferon-beta 1b (Betaseron)
- 2: MS patients or patients with CIS(Clinically isolated syndrome)who decided to postpone the treatment with IFN-beta

INTERVENTIONS:
Drug: Interferon-beta 1b (Betaseron) — Treatment of patients with FDA-approved Rx
  Groups: 1

SUMMARY:
The purpose of this study is to determine whether interferon-beta impairs the ability of plasmacytoid dendritic cells to promote pathogenic immune responses in patients with multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 to 60 year old, inclusive.
* Diagnosis of a relapsing form of multiple sclerosis as determined by revised McDonald Criteria or at least one clinical demyelinating episode with abnormal brain MRI study based on CHAMPS criteria
* Expanded disability status scale (EDSS) score less than 6 at entry.
* Understand and sign written informed consent prior to any testing under this protocol, including screening tests and evaluations that are not considered part of the subject's routine care.

Exclusion Criteria:

* Treatment with corticosteroids within one month prior to the study. Treatment with immunomodulatory drugs within last 3 months prior to the study.
* No history of treatment with Interferon-beta(IFN-beta) based drugs to exclude the possibility of IFN-beta neutralizing antibodies
* Any patient who is pregnant, intend to become pregnant, or breastfeeding at any time of the study.
* History of any significant cardiac, gastrointestinal, hepatic, pulmonary, or renal disease; immune deficiency; or other medical conditions that would preclude IFN-beta therapy.
* Primary Progressive Multiple Sclerosis patients or patients with Secondary Progressive Multiple Sclerosis with lack of recent clinical relapses for more than 2 years

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Multiple Sclerosis Clinic patient
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2007-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Relative gene expression in plasmacytoid dendritic cells (pDCs) | Change in gene expression in 12 weeks
  Gene expression is tested in pDCs separetd from peripheral blood of human subjects at baseline and at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin Balashov, M.D., Ph.D., Principal Investigator — Rutgers Robert Wood Johnson Medical School
Locations (1):
- Rutgers-RWJMS, New Brunswick, New Jersey, United States

REFERENCES:
- [Background] Aung LL, Brooks A, Greenberg SA, Rosenberg ML, Dhib-Jalbut S, Balashov KE. Multiple sclerosis-linked and interferon-beta-regulated gene expression in plasmacytoid dendritic cells. J Neuroimmunol. 2012 Sep 15;250(1-2):99-105. doi: 10.1016/j.jneuroim.2012.05.013. Epub 2012 Jun 9. PMID 22688425
- [Result] Balashov KE, Aung LL, Vaknin-Dembinsky A, Dhib-Jalbut S, Weiner HL. Interferon-beta inhibits toll-like receptor 9 processing in multiple sclerosis. Ann Neurol. 2010 Dec;68(6):899-906. doi: 10.1002/ana.22136. PMID 21061396
- [Result] Aung LL, Fitzgerald-Bocarsly P, Dhib-Jalbut S, Balashov K. Plasmacytoid dendritic cells in multiple sclerosis: chemokine and chemokine receptor modulation by interferon-beta. J Neuroimmunol. 2010 Sep 14;226(1-2):158-64. doi: 10.1016/j.jneuroim.2010.06.008. PMID 20621365